CLINICAL TRIAL: NCT02503345
Title: A Phase 2b, Multi-center, Randomized, Double Blind, Placebo-controlled, Crossover Study to Evaluate Multiple Doses of ALLN-177 in Recurrent Calcium Oxalate Kidney Stone Formers With Hyperoxaluria
Brief Title: Evaluate the Effect of ALLN-177 in Reducing Urinary Oxalate in Patients With Hyperoxaluria and Kidney Stones
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000649
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2017-01

CONDITIONS: Secondary Hyperoxaluria; Nephrolithiasis; Kidney Stones; Hyperoxaluria; Dietary Hyperoxaluria
Keywords: Kidney Stones; Nephrolithiasis; Urine Oxalate; Hyperoxaluria; Enteric Hyperoxaluria; Idiopathic Hyperoxaluria; Urological Diseases; Kidney Diseases; Dietary Oxalate
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi; Hyperoxaluria; Urologic Diseases; Kidney Diseases | interventions — reloxaliase; oxalate decarboxylase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo capsules (1, 2 or 5) PO TID
  Interventions: Drug: Placebo
- ALLN-177 low dose (Experimental): ALLN-177 1,500 units/meal PO TID
  Interventions: Drug: ALLN-177 low dose
- ALLN-177 mid dose (Experimental): ALLN-177 3,000 units/meal PO TID
  Interventions: Drug: ALLN-177 mid dose
- ALLN-177 high dose (Experimental): ALLN-177 7,500 units/meal PO TID
  Interventions: Drug: ALLN-177 high dose

INTERVENTIONS:
Drug: ALLN-177 low dose — ALLN-177 1,500 units (1 capsule)/meal PO 3 times per day
  Other Names: Oxalate decarboxylase
  Arms: ALLN-177 low dose
Drug: ALLN-177 mid dose — ALLN-177 3,000 units (2 capsules)/meal PO 3 times per day
  Other Names: Oxalate decarboxylase
  Arms: ALLN-177 mid dose
Drug: ALLN-177 high dose — ALLN-177 7,500 units (5 capsules)/meal PO 3 times per day
  Other Names: Oxalate decarboxylase
  Arms: ALLN-177 high dose
Drug: Placebo — Placebo: 1, 2 or 5 capsules with meals PO 3 times per day
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of different doses of ALLN 177 for reducing urinary oxalate excretion in patients with secondary hyperoxaluria and recurrent kidney stones.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo controlled study to evaluate the efficacy of ALLN 177 compared with placebo in reducing the urinary excretion of oxalate in subjects with secondary hyperoxaluria and kidney stones. ALLN-177 is an orally administered form of oxalate decarboxylase. The goal of therapy with ALLN-177 is to reduce urinary oxalate excretion by decreasing the absorption of oxalate from the gastrointestinal tract.

Eligible subjects will be randomized to 7 days of treatment with a dose ALLN-177 or placebo and following a washout period, crossed over to an alternate treatment. Urinary oxalate excretion will be assessed by 24-hr urine collections throughout the study.

The study allows for up to 60 subjects.

ELIGIBILITY:
Inclusion Criteria:

* History of enteric or idiopathic hyperoxaluria and at least one kidney stone within the past 2 years
* Hyperoxaluria at screening
* May be taking drugs for the prevention of stone disease

Exclusion Criteria:

* Hyperuricosuria
* Glomerular filtration rate < 55 mL/min/1.73m2
* Hypercalcemia or hypothyroidism
* Obstructive uropathy, chronic urosepsis, renal failure, renal tubular acidosis, primary hyperparathyroidism, primary hyperoxaluria, pure uric acid and cystine stones, and/or medullary sponge kidney
* Treatment with cholestyramine
* Average daily dietary intake of oxalate <75 mg per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mean urinary oxalate excretion (mg/24 h) following treatment | on 7 days of treatment

SECONDARY OUTCOMES:
Change from baseline in mean urinary oxalate excretion (mg/24 h) | on 7 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Kausz, MD MS, Study Director — VP Clinical Development
Locations (16):
- United States (16):
  - Tower Urology, Los Angeles, California
  - Atlantic Urological Associates, Daytona Beach, Florida
  - Mayo Clinic - Nephrology And Hypertension, Jacksonville, Florida
  - Northwestern Feinberg School Of Medicine - Urology Department, Chicago, Illinois
  - IU Health Physicians Urology, Indianapolis, Indiana
  - Anne Arundel Urology, Annapolis, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Brooklyn Urology Research Group, Brooklyn, New York
  - North Shore Long Island Jewish Health System/The Arthur Miller Institute for Urology, Lake Success, New York
  - New York University - Division Of Nephrology, New York, New York
  - The Urology Group, Cincinnati, Ohio
  - Cleveland Clinic-Urology, Cleveland, Ohio
  - Omega Clinical Research, Warwick, Rhode Island
  - UT Southwestern Medical Center - Urology, Dallas, Texas
  - Urology of Virginia, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No